CLINICAL TRIAL: NCT06555796
Title: A Phase 1b, Open-label, Multicenter Study Evaluating the Safety, Tolerability, and Efficacy of Xaluritamig in Subjects With High-risk Biochemical Recurrence of Nonmetastatic Castration-sensitive Prostate Cancer After Definitive Therapy
Brief Title: Evaluation of Xaluritamig in High-Risk, Biochemically Recurrent, Non-metastatic Castrate-sensitive Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230238
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer; High-risk Biochemical Recurrence; High Risk Biochemical Recurrence of Non-metastatic Castration-sensitive Prostate Cancer; Non-metastatic Castration-sensitive Prostate Cancer
Keywords: Xaluritamig; T-Cell Engager; AMG509; STEAP1; Immunotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Xaluritamig (Experimental): Xaluritamig will be administered as a short-term intravenous (IV) infusion for a total of 6 cycles. One treatment cycle consists of 28 days for cycles 1-2 and 56 days for cycles 3-6.
  Interventions: Drug: Xaluritamig

INTERVENTIONS:
Drug: Xaluritamig — IV infusion
  Other Names: AMG 509

SUMMARY:
The main objective of this study is to evaluate the safety and tolerability of xaluritamig monotherapy in adult participants with high-risk biochemical recurrent (BCR) nonmetastatic castration-sensitive prostate cancer (nmCSPC).

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed adenocarcinoma of the prostate at initial biopsy, without neuroendocrine differentiation, signet cell, or small cell features.
* Prostate cancer initially treated by radical prostatectomy (RP) or radiotherapy (XRT) (including brachytherapy) or both (eg, salvage radiotherapy), with curative intent.
* PSA doubling time ≤ 12 months.
* Participants must have biochemically recurrent disease after definitive treatment to prostate by either RP or XRT.
* Screening PSA by the local laboratory ≥ 0.2 ng/mL for participants who had RP (with or without XRT) as primary treatment for prostate cancer or at least 2 ng/mL above the nadir (local assessments) for participants who had XRT or brachytherapy only as primary treatment for prostate cancer.
* Serum testosterone ≥ 150 ng/dL (5.2 nmol/L).
* Participants must have undergone a prostate-specific membrane antigen (PSMA) positron emission tomography (PET) scan during or within 3 months of screening.

Exclusion Criteria

* Present evidence of metastatic disease in conventional CT scan and/or bone scan
* Participants that present PSMA-positive lesions in the PSMA PET scan may be enrolled if the conventional imaging does not show suspicion of metastatic disease.
* Prior hormonal therapy, exceptions include:

  * Neoadjuvant/adjuvant therapy to treat prostate cancer ≤ 36 months in duration and ≥ 9 months before enrollment, or
  * A single dose or a short course (≤ 6 months) of hormonal therapy given for rising PSA ≥ 9 months before enrollment.
* Prior cytotoxic chemotherapy, aminoglutethimide, ketoconazole, abiraterone acetate, enzalutamide, apalutamide, or darolutamide for prostate cancer.
* Abiraterone acetate, enzalutamide, apalutamide, or darolutamide are allowed if administered in a neoadjuvant/adjuvant setting ≤ 36 months in duration and ≥ 9 months before enrollment.
* Prior systemic biologic therapy, including immunotherapy, for prostate cancer.
* If, in the investigator's opinion, salvage therapy is the preferred intervention.
* Autoimmune disease requiring systemic immunosuppression within the past 2 years.
* Participant with symptoms and/or clinical signs and/or radiographic signs that indicate an acute and/or uncontrolled active systemic infection within 7 days prior to the first dose of study treatment.
* Requirement for chronic systemic corticosteroid therapy (prednisone dose > 10 mg/day or equivalent) or any other immunosuppressive therapies (including anti tumor necrosis factor alpha [TNFα] therapies) unless stopped (with adequate tapering) within 7 days prior to dosing.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-10-08 (Estimated); Study Completion 2028-12-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to approximately 2 years
  Events categorized as adverse events (AEs) starting on or after first dose of investigational product (xaluritamig) as determined by the flag indicating if the AE started prior to the first dose on the Events Electronic Case Report Form (eCRF) and including 30 days after the last dose of investigational product (xaluritamig) or end of study date, whichever is earlier.
Number of Participants Experiencing Treatment-related Adverse Events (TRAEs) | Up to approximately 2 years
  A TRAE is any TEAE that per investigators' review has a reasonable possibility of being caused by the investigational product (xaluritamig) determined by the flag indicating an event may have been caused by the investigational product (xaluritamig) on the Events eCRF. In the unlikely event that the flag is missing, the TEAE will be considered related.

SECONDARY OUTCOMES:
Time to Prostate-specific Antigen (PSA) Progression | Up to 50 months
Number of Participants With a PSA 50 Response | Up to approximately 50 months
Number of Participants With a PSA 90 Response | Up to approximately 50 months
Duration of PSA 50 Response | Up to approximately 50 months
Duration of PSA 90 Response | Up to approximately 50 months
Number of Participants With Undetectable PSA | Up to approximately 50 months
Time to Initiation of Androgen Deprivation Therapy or Androgen Receptor Directed Therapy | Up to approximately 50 months
Time to First use of new Anticancer Therapy | Up to approximately 50 months
Time to Metastatic Disease/Progression | Up to approximately 50 months
Metastasis-free Survival (MFS) | Up to approximately 50 months
Number of Participants Completing Xaluritamig Monotherapy Treatment | Up to approximately 24 months
Maximum Serum Concentration (Cmax) of Xaluritamig | Up to approximately 24 months
Time to Cmax (Tmax) of Xaluritamig | Up to approximately 24 months
Area Under the Concentration-time Curve (AUC) Over the Dosing Interval of Xaluritamig | Up to approximately 24 months
Terminal Half-life (t1/2) of Xaluritamig | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- United States (8):
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Levine Cancer Institute, Charlotte, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (3):
  - Chris OBrien Lifehouse, Camperdown, New South Wales
  - Cabrini Hospital, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com